CLINICAL TRIAL: NCT03314038
Title: Validating Features of Traditional Chinese Syndrome Patterns for Chronic Atrophic Gastritis Malignant Transformation: A Cross-sectional Study
Brief Title: Syndrome Patterns for Chronic Atrophic Gastritis Malignant Transformation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing University of Chinese Medicine (Other)
Collaborators: The University of Science and Technology of China (Other); China Academy of Chinese Medical Sciences (Other); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Dr. Xia Ding, Professor, Beijing University of Chinese Medicine
Other Study IDs: 81630080-CAG-CS
Record Dates: First submitted 2017-10-15; First posted 2017-10-19 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: TCM Syndrome of Chronic Atrophic Gastritis
Keywords: Chronic Atrophic Gastritis; Malignant Transformation; Syndrome; Traditional Chinese Medicine; Cross-sectional Study
MeSH Terms: conditions — Gastritis, Atrophic; Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and gastric mocusa tissue sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic atrophic gastritis (CAG) is acknowledged as the precancerous stage of gastric cancer (GC). The present study aims to explore Traditional Chinese Medicine (TCM) syndrome features in different stages of CAG malignant transformation respectively. The proposed study is a cross-sectional study based participant survey conducted in 4 hospitals in Beijing, China. After obtaining informed consent, a total of 2000 study patients will be recruited on-site in hospitals.

DETAILED DESCRIPTION:
CAG is acknowledged as the precancerous stage GC. Active treatment of CAG is vital in arresting malignant transformation. Traditional Chinese medicine (TCM) has been widely used in treating CAG and preventing GC in China. To date, few study has been conducted to assess the syndrome features of different stages of CAG malignant transformation combining TCM indicators.

The present study aims to explore TCM syndrome features in different stages of CAG malignant transformation. The proposed study is a registry study based participant survey conducted in 4 hospitals in Beijing, China. After obtaining informed consent, a total of 2000 eligible study patients will berecruited on-site in hospitals.

Comparative analysis of prevalence of presenting TCM features is conducted using frequency analysis and chi-squared tests, and expressed with composition ratios. Exploratory factor analysis,correspondence analysis, association rule analysis, hierarchical clustering analysis, and complex system entropy clustering analysis will be performed respectively for validating features of syndrome in different stages of CAG malignant transformation.

Previous reports on TCM syndrome features for CAG exist, but no studies have been undertaken base on large-sampled study design and detailed analysis in different stages of CAG malignant transformation respectively.

The outcome of our study has the potential to clerify core TCM pathogenesis of CAG, facilitate early intervention, and promote optimization of treatment strategies of CAG malignant transformation by TCM.

ELIGIBILITY:
Inclusion Criteria:

* (1) 18-75 years of age; (2) Meeting diagnostic criteria of CAG after upper gastrointestinal endoscopy; (3) Willing to cooperate with data, tissue sample, and blood sample collection during recruitment; (4) Willing to respond truthfully and timely to researcher queries after recruitment, able to cooperate with data, tissue sample and blood sample collection during follow-ups; (5) Willing to sign informed consent.

Exclusion Criteria:

* (1) Meeting past history of previous stomach surgery; (2) Unable to participate in data, tissue sample or blood sample collection for any reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a multicenter cross-sectional study conducted in 4 hopitals in Beijing, China,lleaded by Beijing University of Chinese Medicine. According to the inclusion and exclusion criteria, 2000 eligible participants will be involved in this study.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
TCM syndrome | one time at involvement (1 day)
  According to the symptoms and physical signs of patients to determine the syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Xia Ding, MD, Principal Investigator — Beijing University of Chinese Medicine
Locations (1):
- Beijing University of Chinese Medicine, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhang Y, Liu Y, Song R, Zhang L, Su Z, Li Y, Chen R, Shi N, Zhao X, Du S, Ding X. Validating traditional Chinese syndrome features in varied stages of chronic gastritis malignant transformation: study protocol for a cross-sectional study. BMJ Open. 2018 Aug 30;8(8):e020939. doi: 10.1136/bmjopen-2017-020939. PMID 30166291